CLINICAL TRIAL: NCT03700125
Title: Feasibility Study of a Pre-hospital Extra-corporeal Membrane Oxygenation (ECMO) Capable Advanced Resuscitation Team at Achieving Blood Flow Within 30 Minutes in Patients With Refractory Cardiac Arrest.
Brief Title: Pre-hospital ECMO in Advanced Resuscitation in Patients With Refractory Cardiac Arrest. ( SUB30 )
Acronym: SUB30
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Bodychillz Ltd (Industry); Maquet Cardiopulmonary GmbH (Industry); Stryker Nordic (Industry); London's Air Ambulance Charity, Registered Charity (801013) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012543; 244748 (Other: IRAS)
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Death, Sudden, Cardiac; Out-Of-Hospital Cardiac Arrest; Ventricular Fibrillation; Cardiopulmonary Arrest With Successful Resuscitation
Keywords: Advanced life support (ALS); Extra-corporeal Membrane Oxygenation Resuscitation (ECMO)
MeSH Terms: conditions — Death, Sudden, Cardiac; Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Intervention Model Description: Single centre feasibility study of a complex intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECMO resuscitation (Experimental): 6 patients who meet the eligibility criteria will be treated by pre-hospital advanced physician/ paramedic cardiac arrest team that is ECMO capable and can establish ECMO flow within 30 minutes of collapse
  Interventions: Procedure: ECMO resuscitation

INTERVENTIONS:
Procedure: ECMO resuscitation — Extracorporeal Cardio-Pulmonary Resuscitation (ECPR) using ECMO within 30 minutes of cardiac arrest
  Other Names: Extracorporeal Membrane Oxygenation

SUMMARY:
To establish whether a pre-hospital advanced physician/ paramedic cardiac arrest team that is ECMO capable can establish ECMO flow within 30 minutes of collapse. The Sub30 study will investigate the technical and logistical feasibility of instituting pre-hospital Extracorporeal Cardiopulmonary Resuscitation (ECPR) within 30 minutes of collapse for selected patients (n=6) in a geographical sector of Greater London. It will achieve this through a unique collaboration between the primary emergency dispatch and response services (London Ambulance Service NHS Trust, LAS), pre-hospital practitioners (LAS and London Air Ambulance) and clinicians in ECMO (Barts Health NHS Trust).

DETAILED DESCRIPTION:
Every year, in London, the ambulance service treats over 4,000 patients who have a had a cardiac arrest (or their heart has stopped). Less than 1 in 10 patients survive to get home. Some of those who survive have severe brain damage since their brains did not receive blood and oxygen when their heart was stopped. The ambulance service in London manages to get to a patient, on average, 7 minutes following a 999 call. The paramedics are very skilled in restarting people's hearts and often manage this in less than 10 minutes. However, sometimes it can take much longer or not be possible. The risks of a patient dying or suffering brain damage increase the longer it takes to restart the heart, particularly after about 20-30 minutes. An extracorporeal membrane oxygenation (ECMO) machine may reduce these risks by pumping a patient's blood through an artificial lung and to their vital body organs - temporarily replacing the function of the heart and lungs. The ECMO is used in normal care to support patients after a cardiac arrest once a patient reaches the hospital, but in this study we want to see if the ECMO can be used very soon after the cardiac arrest is reported via the 999 call.

In the Sub30 study, the ECMO team and machine to travel immediately to where the patient collapses rather than wait for the patient to be moved to a hospital. The study hypothesis is that the ECMO will be started faster and that this may improve patient survival and outcomes.

The ECMO team consists of three senior doctors and a paramedic. They attend patients who have collapsed and start ECMO if standard advanced resuscitation techniques fail to restart the heart in 20 minutes. The team will aim to have the ECMO machine started within 30 minutes of the 999 call. The team have achieved this in training and the current study will assess whether it is possible to do this in six patients in real-life.

A target of thirty minutes to achieve ECMO flow or return of spontaneous circulation (ROSC) is less than in published series to date. This can be achieved by:

* integration into an established pre-hospital emergency response services that aggressively pursue ROSC through optimised Advanced Life Support
* immediate deployment of an ECPR-capable cardiac arrest team as a primary resource, as opposed to delayed secondary deployment. Dispatch will be done by the established Advanced Paramedic Practitioner (APP) desk of London Ambulance Service, with the objective to reach the patient within 8-10 minutes of the 999 call.
* early placement of guide-wires into the femoral vessels during on-going conventional CPR, a procedure with low complication risk that does not commit the team to ECPR but will minimise the delay to ECPR support if conventional resuscitative techniques are not successful within 20 minutes
* facilitated guide-wire placement through real-time wireless ultrasound delivered to the operator through augmented reality smart glasses.

Some out of hospital cardiac arrests (OHCA) are irreversible in nature and ECPR would not provide benefit to these patients. The ECPR team will not be task fixated on providing ECPR, but also supportive of the APP primary responders and provide ECPR only in settings of refractory cardiac arrest that fulfils the study criteria, that have been chosen based on best available evidence to identify those patients in whom ECPR is likely to be of benefit.

If pre-hospital ECMO is feasible within 30 minutes of chest compressions starting, then a larger randomised controlled study of clinical and cost effectiveness is merited. Optimisation of the delivery of ECPR is vital, prior to a controlled study, in order to maximise any potential benefits for patients.

Data from Sub30 will inform the design of such studies enabling an estimation of the size of any potential outcome benefits and the likely affordability for a healthcare service.

ELIGIBILITY:
Inclusion Criteria:

Adult patients who:

* have a witnessed out-of-hospital cardiac arrest
* a presumed cardiac aetiology to their cardiac arrest
* receive bystander chest compressions within 3 minutes
* remain in cardiac arrest at 20 minutes following the call to the emergency services or fail to sustain ROSC in the pre-hospital setting

Exclusion Criteria:

The following patients will not be suitable for entry into the study:

* Known to be are visibly appear younger than 18 years old or older than 65 years.
* Known or visible advanced pregnancy (when resuscitative hysterotomy should be performed)
* No signs of life (physical movement or breathing) AND evidence of ineffective chest compressions suggested by:
* absence of electrical activity at 20 minutes time out OR
* end tidal carbon dioxide level of less than 1.3 kPa (10 mmHg)
* Evidence from others present at the scene or patient examination that ECMO unlikely to benefit patient (e.g. advanced malignancy, severe frailty).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Finney, Principal Investigator — Barts & The London NHS Trust
Locations (2):
- United Kingdom (2):
  - St Bartholomew's Hospital, London
  - London Ambulance Service Trust, London

IPD SHARING:
Plan to Share IPD: No
There is no plan to share study participant data

REFERENCES:
- [Background] Singer B, Reynolds JC, Davies GE, Wrigley F, Whitbread M, Faulkner M, O'Brien B, Proudfoot AG, Mathur A, Evens T, Field J, Monk V, Finney SJ; International ECMO Network (ECMONet). Sub30: Protocol for the Sub30 feasibility study of a pre-hospital Extracorporeal membrane oxygenation (ECMO) capable advanced resuscitation team at achieving blood flow within 30 min in patients with refractory out-of-hospital cardiac arrest. Resusc Plus. 2020 Dec;4:100029. doi: 10.1016/j.resplu.2020.100029. Epub 2020 Oct 8. PMID 33403364
- [Result] Singer B, Hla TTW, Abu-Habsa M, Davies G, Wrigley F, Faulkner M, Finney SJ. Sub30: Feasibility study of a pre-hospital extracorporeal membrane oxygenation (ECMO) in patients with refractory out-of-hospital cardiac arrest in London, United Kingdom. Resuscitation. 2025 Feb;207:110455. doi: 10.1016/j.resuscitation.2024.110455. Epub 2024 Dec 5. PMID 39645021

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ECMO Resuscitation
Started | 5 (Study stopped prior to recruitment of final patient as medical device had a temporary suspension of its CE license. This was considered to not impact on the results of this feasibility study.)
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Successfully Established With Pre-hospital ECPR
Description: The primary endpoint is the proportion of patients successfully established with pre-hospital ECPR within 30 minutes of collapse
Time Frame: Within 30 minutes of collapse
Measure: Count of Participants; unit: Participants
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Ambulance Dispatch
Description: Number of patients not dispatched to as travel time too great/team unavailable
Time Frame: Within 30 minutes of collapse
Population: The ambulance dispatch centre is very busy with always many calls waiting to be answered. If calls were not within criteria (not cardiac arrests, not suitable, too far away) the call operators moved on to the next call and did not record a non-activation. As the operators did not record the non-activation, it was not feasible to collect these data
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 0

3. Secondary Outcome: Successful Cannulation
Description: The number of patients successfully cannulated 31 and 45 minutes
Time Frame: between 31 and 45 minutes; and 46 and 60 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
Participants | 2

4. Secondary Outcome: Number of Patients With Return of Spontaneous Circulations (ROSC)
Description: The number of patients patients who achieve ROSC prior to the 20 minutes timeout, number of patients in refractory cardiac arrest at 20 minutes in whom ROSC is achieved prior to ECMO flow
Time Frame: Within 20 minutes of cardiac arrest
Measure: Count of Participants; unit: Participants
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Emergency Call-out Time Frame
Description: The time interval between call to the emergency services and ECPR team arrival
Time Frame: At 30 minutes after cardiac arrest
Measure: Median (Full Range); unit: Minutes
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
Minutes | 16 [5 to 22]

6. Secondary Outcome: Successful Guide Wire Placement
Description: The proportion of potentially supportable patients in whom guidewire placement is attempted and achieved
Time Frame: Up to 30 minutes after cardiac arrest
Measure: Count of Participants; unit: Participants
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
Participants | 5

7. Secondary Outcome: Incidence of ECPR-related Complications
Description: Assessment of ECPR-related complications, such as incidence of vascular damage, haemorrhage requiring transfusion and new organ dysfunction
Time Frame: Duration of ECMO run, between 3 - 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
Participants
  Limb ischaemia | 1
  Cannulation site bleeding | 1
  Microbubbles in right heart | 1
  No ECPR serios event | 2

8. Secondary Outcome: Clinical Outcome Via FIM at 3 Months
Description: Assessment of functional status at hospital discharge using the Functional Independence Measure - FIM (18 item scale, measure of dependence. The higher the score, the more independent the patient is in performing the task).
Time Frame: 3 months
Population: 3 patients died and could not be assessed. Remaining 2 patients were no longer in hospital at the planned assessment time. The study team lacked the resource to assess at alternative centres and this feasibility study demonstrated that this measure is complex to collect. Noted as protocol variations.
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 0

9. Secondary Outcome: Clinical Outcome Via MRS at 3 Months
Description: Assessment of functional status at hospital discharge using the modified Rankin Scale (MRS) (scale 0-6, measuring the degree of disability or dependence in the daily activities, where 0 is no symptoms and 6 is dead)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
Participants
  0 | 0
  1 | 0
  2 | 0
  3 | 0
  4 | 1
  5 | 1
  6 | 3

10. Secondary Outcome: Duration of Hospital Stay (ICU)
Description: Assessment of health resources used for the duration of Intensive Care Unit stay
Time Frame: 1-3 months
Measure: Median (Full Range); unit: days
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 5
days | 16 [2 to 25]

11. Secondary Outcome: Number of Acute Hospital Admissions Post Discharge
Description: Assessment of health resources used for further hospital admissions following discharge.
Time Frame: 3 months
Measure: Median (Full Range); unit: admissions post discharge
Arm/Group | ECMO Resuscitation
Number analyzed (Participants) | 2
admissions post discharge | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 90 days after study entry
Arm/Group | ECMO Resuscitation
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECMO Resuscitation (N=5)
Limb ischaemia (Cardiac disorders) | 1 (1)
Microbubbles in right heart on echo (Cardiac disorders) | 1 (1)
Cannulation site bleeding (Vascular disorders) | 1 (1)
Calibration error on ECMO machine (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECMO Resuscitation (N=5)
Haemoperitoneum/Haemomediastinum (Cardiac disorders) | 1 (1)
Bleeding following IABP removal (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT03700125/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03700125/SAP_001.pdf